CLINICAL TRIAL: NCT03388931
Title: Radiotherapy Dose Escalation in Locally Advanced Squamous Cell Carcinoma of the Larynx or Hypopharynx
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of subject enrollment
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702707; OCR17025 (Other: UF OnCore)
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Advanced Squamous Cell Carcinoma
Keywords: Radiotherapy Dose Escalation
MeSH Terms: interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): Increased dose of radiation therapy for locally advanced squamous cell carcinoma of the larynx or hypopharynx. Patients will also receive standard-of-care chemotherapy with the treatment regimen to be determined by the treating physicians.
  Interventions: Radiation: Radiation Therapy; Combination Product: Chemotherapy

INTERVENTIONS:
Radiation: Radiation Therapy — Increased radiation therapy dose
Combination Product: Chemotherapy — Standard-of-care chemotherapy with treatment regimen to be determined by the treating physician

SUMMARY:
This is a phase 2 single arm study of a novel schedule of hyperfractionated radiotherapy (RT) in combination with our standard chemotherapy program for patients with stage 3-4 squamous cell carcinoma of the larynx. The primary hypothesis of our study is that the study program will improve Laryngectomy-Free Survival compared to historical controls. The study is limited to patients who would be receiving primary RT-C as standard therapy off-study.

DETAILED DESCRIPTION:
The novel radiotherapy schedule that is the subject of this study is only slightly different from the program that has been used in the cooperative group trial RTOG 9003. The radiation therapy dose schedule in our study twice-daily alternating fractions over 30 treatment days. The Biologically Effective Dose (BED) of this schedule is about 11% higher than our standard schedule twice-a-day. During radiotherapy, patients will receive chemotherapy with our standard program of weekly.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age (no upper age limit)
* Biopsy proven squamous cell carcinoma of the glottis or supraglottic larynx or hypopharynx with the following T,N and M stages:
* Glottic Larynx:

T3-4: Any primary tumor volume

* Supraglottic Larynx:

T2: Primary tumor volume > 4.0cc T3-4: Any primary tumor volume

* Hypopharynx:

T2: Primary tumor volume > 4.0cc T3-4: Any primary tumor volume

* N-Stages (the same for all primary sites): All N-stages
* M-Stages (the same for all primary sites): M0 or M1suitable for curative attempt with Stereotactic Body Radiation Therapy.
* Radiologic evaluation of the chest within 12 weeks prior to treatment; at a minimum, chest x-ray is required. CT imaging of the chest or PET/CT is acceptable.
* ECOG Performance Status 0-2
* CBC/differential obtained within 8 weeks prior to treatment, with adequate bone marrow function defined as follows:
* Platelets ≥ 100,000 cells/mm3
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
* Adequate renal and hepatic function within 4 weeks prior to treatment, defined as follows:
* Serum creatinine < 2.0 mg/dl
* Total bilirubin < 2 x the institutional ULN
* AST or ALT < 3 x the institutional ULN.

  *Note that physician attestation of patient having no known history of liver disease can take the place of bilirubin and AST/ALT labs.
* Negative pregnancy test within 2 weeks prior to treatment for women of childbearing potential
* Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment and for 6 weeks following treatment.
* Patients must be deemed able to comply with the treatment plan and follow-up schedule.
* Patients must provide study specific informed consent prior to study entry

Exclusion Criteria:

* Prior history of radiation therapy to the head and neck that would likely increase the risk of serious complications from the RT delivered on this protocol
* Prior history of head and neck cancer with the exception of nonmelanoma skin cancer.
* Currently taking Disease Modifying Rheumatoid Drugs (DMRDs)
* Severe, active co-morbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; Note, however, coagulation parameters are not required for entry into this protocol.
* Pre-existing ≥ grade 2 neuropathy
* Prior organ transplant
* Systemic lupus
* Psoriatic arthritis.
* Known HIV positive. HIV positive patients are known to have worse clinical outcomes especially for local, regional, and distant cancer control. This poorer prognosis is thought to be secondary to a compromised immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Whether radiation therapy dose escalation as used in our study will improve Laryngectomy-Free Survival compared to historical controls in patients with locally advanced squamous cell carcinoma of the larynx. | Up to 2 years
  Patients will receive an increased dose of radiation therapy

SECONDARY OUTCOMES:
Patient reported quality of life | Up to 2 years
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients Likert scales 1-4,(1 = All, 2 = Little, 3 = a Bit, 4 = Very much)
Psychosocial function | Up to 2 years
  Voice Handicap Index (VHI) a 30-item questionnaire. Likert scale 0- 4, 0 = never and 4 Always) A change between two administrations of 18 points represents a significant shift in psychosocial function.
Swallowing ability. | Up to 2 years
  The MD Anderson Symptom Inventory (MDASI) is a multi-symptom patient-reported outcome (PRO) measure for clinical and research use. Use the MDASI to assess the severity of symptoms experienced by patients with cancer and the interference with daily living caused by these symptoms.MD Anderson Dysphagia Index (MDADI)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amdur, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States